CLINICAL TRIAL: NCT02598700
Title: Measurement and Quantitative Correlation of Spinopelvic Parameters and Acetabular Cup Orientation Between Standing and Sitting to Define a Better Functional Anteversion Safe Zone in Total Hip Arthroplasty
Brief Title: Correlation of Spinopelvic Parameters and Acetabular Cup Orientation
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00066248
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Hip Osteoarthritis; Complications; Arthroplasty
Keywords: total hip arthroplasty; imaging; arthritis; surgical technique
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In total hip arthroplasty, cup anteversion is an important factor in stability. Lewinnek's safe zone and functional anteversion are often used to assess appropriate orientation. However, these approaches do not consider the effect of the spinopelvic chain and lumbar mobility when in the seated position. This study will measure functional anteversion when standing and sitting with patient-specific computer models and define a quantitative relationship between the change in functional anteversion and spinopelvic parameters. This will challenge the historical paradigm of the safe zone and provide a tool to define anteversion based on a patient's mechanics and reduce risk of dislocation.

DETAILED DESCRIPTION:
In total hip arthroplasty (THA), incorrect cup orientation markedly increases the risk of dislocation, wear, and impingement. The primary method of cup placement is based on the surgeon's interpretation of orientation within a "safe zone" defined by Lewinnek almost 40 years ago. This approach has undergone little change despite consistent dislocation rates and a large proportion of dislocations occurring in patients with cups within the safe zone. One reason for this may be that it does not account for a patient's natural pelvic posture, which affects the functional cup anteversion. Some modern techniques of cup placement assess a functional anteversion based on supine and others on standing orientation. However, these methods do not account for lumbar mobility and the effects on spinopelvic mechanics when in the seated position, the most common position in which dislocation occurs. The investigators have shown that patients with lumbar fusion have a higher rate of THA dislocation. This risk also correlated with length of fusion construct. This suggests that decreased lumbar mobility, whether a result of arthrodesis, disease or age related degeneration, may play an important role in the risk of THA dislocation. Some studies have measured change in pelvic orientation and cup anteversion between sitting and standing. Others have used modeling to estimate change in functional anteversion based on pelvic tilt. Presently, however, there are no studies that have investigated the quantitative relationship, in vivo, between patient-specific changes in spinopelvic parameters and cup anteversion between sitting and standing. Within this exploration, identification of an appropriate safe zone in individuals with mobility restrictions of the lumbar spine is not possible.

The investigators will test the hypothesis by addressing the aims presented below. These aims will be approached by directly measuring the spinopelvic parameters on standing and seated radiographs in 100 patients who have undergone primary THA. Computer models of cups and pelvises generated from patient-specific pelvis CTs will be manipulated based on the measured changes in pelvic alignment. The change in functional cup anteversion will then be directly measured from each patient's model.

Specific Aim #1: To quantify the relationship between the change in pelvic tilt and functional acetabular cup anteversion between the standing and sitting positions in patients who have undergone primary THA. The investigators hypothesize that there will be a directly proportional relationship between the increase in pelvic tilt and increase in functional anteversion. The investigators anticipate that Aim #1 will identify the importance of functional anteversion in the seated position and support its consideration when defining a patient-specific cup safe zone. This data will serve as the foundation for development of a clinical tool used in pre-operative planning and post- operative rehabilitation that accounts for spinopelvic mechanics to maintain safe cup orientation when in the vulnerable seated position.

Specific Aim #2: To quantify the relationship between the change in lumbar lordosis and functional acetabular cup anteversion between the standing and sitting positions in patients who have undergone primary THA. The investigators hypothesize that there will be a directly proportional relationship between the decrease in lumbar lordosis and increase in functional anteversion and that patients with history of lumbar immobility will have decreased change in functional anteversion. The data obtained in Aim #2 can be used to identify those at increased risk of dislocation. It will also provide insight into, and a basis for further study of, the relationship between seated functional anteversion and specific etiologies of lumbar immobility (spinal fusion, ankylosing spondylitis, flat back syndrome, degenerative changes, etc.) that may affect THA dislocation.

The overall objective of this study is to define a clinically relevant and applicable quantitative correlation between the change in spinopelvic parameters and change in functional anteversion between the standing and seated positions and challenge the historical safe zone paradigm. The central hypothesis is that the change spinopelvic mobility correlates with the change in functional anteversion. The investigators believe that this quantitative relationship will provide the clinician a tool to identify at-risk THA candidates and make appropriate patient-specific modifications to cup anteversion and post-operative rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

-All patients who have undergone THA with the appropriate pre-operative CT for planning and those who are candidates for primary THA for osteoarthritis will be contacted for recruitment.

Exclusion Criteria:

* inflammatory arthritis
* neuromuscular disorders
* revision surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone THA with the appropriate pre-operative CT for planning and those who are candidates for primary THA for osteoarthritis will be contacted for recruitment. Those with inflammatory arthritides or neuromuscular disorders will not be eligible for the study. Women of childbearing age will also be excluded from this study. Base on the power analysis below, the investigators anticipate eighty-four (84) patients will be enrolled into this study.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Quantitative correlation between change functional anteversion and change in pelvic tilt using patient-specific measurements and computer models. | 1 year
  A quantitative relationship will be generated correlating change in cup anteversion (change in degrees) to change in pelvic tilt (change in degrees) at given inclinations (degrees) as simulated in the model. Statistical analysis will then be performed. Significance of changes between standing and sitting in pelvic tilt and cup anteversion will be assessed with t-test or non-parametric equivalent if appropriate with significance p<0.05. The effect of change in pelvic tilt on change in functional anteversion will be tested using a two-tailed Pearson product moment.
Quantitative correlation between change functional anteversion and change in lumbar lordosis using patient-specific measurements and computer models. | 1 year
  A quantitative relationship will be generated correlating change in cup anteversion (change in degrees) to change in lumbar lordosis (change in degrees). Statistical analysis will then be performed. Significance of changes between standing and sitting in lumbar lordosis and cup anteversion will be assessed with t-test or non-parametric equivalent if appropriate with significance p<0.05. The effect of change in lumbar lordosis on change in functional anteversion will be tested using a two-tailed Pearson product moment.

SECONDARY OUTCOMES:
Presence of lumbar pathology | 1 year
  degenerative disc disease, posterior degenerative disease, osteophytosis, ankylosing spondylitis, scoliosis, or flat back syndrome
Previous lumbar surgery - fusion type | 1 year
  posterior, anterior, or combined
Previous lumbar surgery - length of fusion | 1 year
  number of fusion levels
Total hip arthroplasty dislocation | 1 year
  presence of dislocation
Other total hip arthroplasty complication | 1 year
  loosening, fracture, or infection

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Seyler, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States